CLINICAL TRIAL: NCT00522847
Title: Biochemical Factors for a Dry Eyed Population
Acronym: GARNET
Status: Completed | Type: Observational
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Craig Woods, Research Manager, CCLR
Other Study IDs: P/263/07/L
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Dry Eye
Keywords: Postmenopausal; non dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tears
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare various symptoms and signs of dry-eye as well as stratify characteristics of the tear film in a group of dry-eyed individuals in comparison to a group of non-dry-eyed people. Dry-eye is a condition that significantly impacts the quality of life of the sufferer. These are people who are predominantly female and in the older age groups. Determining what characterises a person with dry-eyes is of importance to understanding the disease process.

DETAILED DESCRIPTION:
Dry eye is a multifactorial disease that results in a wide variety of signs and symptoms, which are often poorly correlated. Recent work has shown that not only are there changes in the composition of the tear film (including cytokines and the presence of various mucin species and tear film proteins) but also quantifiable changes in both the structure and function of the ocular surface, including corneal sensitivity and the appearance of the epithelial cells and the sub-basal neural network. To-date, no published study has attempted to correlate various clinical and morphological changes found in dry eye with tear film and ocular surface biomarkers.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study, for the dry eye group or control, if she:

1. Is Caucasian, and has full legal capacity to volunteer.
2. Is post-menopausal, with menses ceasing more than 12 months ago.
3. Has moderate or severe dry eye symptoms based on dry eye questionnaire and half of the time wants to use eye drops for dry eye symptoms (dry eye group)
4. Has read, understood and signed an information consent letter.
5. Is willing and able to follow instructions and maintain the appointment schedule.
6. Has clear corneas and no active ocular disease.
7. Has had an ocular examination in the last two years.

Exclusion Criteria:

1. Is on hormone replacement therapy (HRT).
2. Ceased menses due to autoimmune disorders, mumps, chemotherapy, pelvic irradiation or smoking.
3. Has rheumatoid arthritis, diabetes, Sjogren's syndrome or any other systemic disease affecting ocular health.
4. Is using any systemic or topical medications (other than eye drops for dry eye symptoms) that may affect ocular health and neuroendocrine system function.
5. Has undergone corneal refractive surgery.
6. Is aphakic.
7. Has any active ocular disease.
8. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study.
9. Is participating in any other type of clinical or research study.
10. Is a contact lens wearer.
11. Has blepharitis.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Fonn, M.Optom, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Contact Lens Research, School of Optometry, Waterloo, Ontario, Canada